CLINICAL TRIAL: NCT07191275
Title: The Effect of TMS on Emotional Valence Evaluation of Aversive Pictures
Brief Title: Study on the Effect of Transcranial Magnetic Stimulation on the Perception of Emotional Images
Acronym: SAME-M
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dominique de Quervain, MD (Other)
Responsible Party: Sponsor-Investigator, Prof. Dominique de Quervain, MD, Director Division of Cognitive Neuroscience, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2025-01622
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Emotional Memory
Keywords: memory; emotional memory; transcranial magnetic stimulation; emotional valence; emotional arousal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants starting with experimental condition (Experimental): Bilateral continuous theta burst stimulation (cTBS) 30 Hz to the temporo-occipital cortex
  Interventions: Device: Experimental continuous 30 Hz thetaburst transcranial magnetic stimulation; Device: Control continuous 30 Hz thetaburst transcranial magnetic stimulation
- Participants starting with control condition (Active Comparator): Active control condition using bilateral continuous theta burst stimulation (cTBS) 30 Hz to the superior parietal cortex
  Interventions: Device: Experimental continuous 30 Hz thetaburst transcranial magnetic stimulation; Device: Control continuous 30 Hz thetaburst transcranial magnetic stimulation

INTERVENTIONS:
Device: Experimental continuous 30 Hz thetaburst transcranial magnetic stimulation — Bilateral continuous theta burst stimulation (cTBS) 30 Hz to the temporo-occipital cortex
  * Frequency: trains of 30 Hz (3 pulses) every 167 ms (frequency of 6 Hz, in the range of theta band)
  * Intensity: 100% of resting motor threshold (rMT)
  * Location: consecutively on left and right temporo-occipital cortex (MNI: -47, -77, 4; 50, -69, -4)
  * Duration: 33.3 seconds for each side
  * Timing: Immediately before showing IAPS pictures (off-line)
  Other Names: cTBS 30Hz; TMS cTBS 30Hz
Device: Control continuous 30 Hz thetaburst transcranial magnetic stimulation — Active control condition using bilateral continuous theta burst stimulation (cTBS) 30 Hz to the superior parietal cortex
  * Frequency: trains of 30 Hz (3 pulses) every 167 ms (frequency of 6 Hz, in the range of theta band)
  * Intensity: 100% of resting motor threshold (rMT)
  * Location: consecutively on left and right superior parietal cortex (MNI: -17, -70, 60; 17, -70, 60)
  * Duration: 33.3 seconds
  * Timing: Immediately before showing IAPS pictures (off-line)
  Other Names: cTBS 30Hz; TMS cTBS 30 Hz

SUMMARY:
The goal of the current clinical trial is to investigate whether transcranial magnetic stimulation (TMS) over specific brain areas can influence the perception of emotional images and emotional memory. TMS is a non-invasive superficial brain stimulation generated by a magnetic field. The results of the study aim to provide valuable insights for the use of TMS in the investigation of mental processes.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* Normotensive (BP 90/60mmHg - 140/90mmHg)
* BMI: 18 - 30 kg/m2
* Fluent in speaking German

Exclusion Criteria:

* Metal in the head area (e.g., splinters, fragments, clips, etc.)
* Implanted neurostimulator (e.g., DBS, epidural/subdural, VNS)
* Cardiac pacemaker or intracardiac lines
* Medication infusion device
* Non removable metal piercings in the head area, pivot teeth (retainers are no exclusion criterion)
* Tattoos (head area) less than 3 months old or older than 20 years
* Condition after neurosurgery
* Hearing problems or tinnitus
* Not able to sit still due to tremor, tics, itching
* History of repeated syncope
* Head trauma diagnosed as concussion or associated with loss of consciousness
* diagnosis of epilepsy, or a convulsion or a seizure in the past of the participant or his/her close family (parents and siblings)
* TMS in the past showing problems
* Spinal or ventricular derivations
* Positive pregnancy test
* Alcohol intake 12 hours before TMS visits
* Regular intake of any medication (excluding oral contraceptives)
* CNS-active medication or illegal drugs 48h before TMS visits
* Individual's rMT above the limits of rTMS device
* Suicidal tendency as measured by Montgomery-Åsberg Depression Rating Scale (MADRS), item 10 > 0

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Emotional valence for aversive pictures | Immediately after the intervention, lasting for approximately 7 minutes
  The mean valence rating of aversive pictures as assessed by a visual analogue scale assessed directly after TMS.

SECONDARY OUTCOMES:
Emotional arousal | Immediately after the intervention, lasting for approximately 7 minutes
  The mean arousal rating of aversive pictures as assessed by a visual analogue scale assessed directly after TMS.
Aversive episodic memory | Approximately one hour after the intervention
  Number of aversive pictures remembered in a free recall pictorial task using IAPS picture set

OTHER OUTCOMES:
Emotional valence for non-aversive pictures | Immediately after the intervention, lasting for approximately 7 minutes
  The mean valence rating of non-aversive pictures as assessed by a visual analogue scale assessed directly after TMS.
Emotional arousal for non-aversive pictures | Immediately after the intervention, lasting for approximately 7 minutes
  The mean arousal rating of non-aversive pictures as assessed by a visual analogue scale assessed directly after TMS.
Non-aversive episodic memory | Approximately one hour after the intervention
  Number of non-aversive pictures remembered in a free recall pictorial task using IAPS picture set

CONTACTS AND LOCATIONS:
Overall Officials: Dominique de Quervain, MD, Principal Investigator — University of Basel, Division of Cognitive Neuroscience
Locations (1):
- University of Basel, Division of Cognitive Neuroscience, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All IPD (de-identified) that underlie results in a publication will be shared upon reasonable request
Access Criteria: All IPD (de-identified) that underlie results in a publication will be shared upon reasonable request for scientific purposes. A reasonable request consists of a short description of the scientific purpose. Requests will be reviewed by the team of the principle investigator.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-20): https://cdn.clinicaltrials.gov/large-docs/75/NCT07191275/Prot_SAP_000.pdf